CLINICAL TRIAL: NCT00921570
Title: The Effects of Renin Angiotensin System Blockage (RAS), Calcium Channel Blocker and Combine Drugs on TWEAK, PTX3 and FMD Levels in Diabetic Proteinuric Patients With Hypertension
Brief Title: The Effects of Renin Angiotensin System Blockage (RAS), Calcium Channel Blocker and Combined Drugs on TWEAK, PTX3 and FMD Levels in Diabetic Proteinuric Patients With Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GATA VALAMEX study
Record Dates: First submitted 2009-06-15; First posted 2009-06-16 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-06

CONDITIONS: Diabetes; Hypertension; Proteinuria
Keywords: TWEAK; FMD; PTX3; Valsartan; Amlodipine; Renin Angiotensin System
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Proteinuria | interventions — Amlodipine; Valsartan

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Amlodipine (Experimental)
  Interventions: Drug: Amlodipine
- Valsartan (Experimental)
  Interventions: Drug: Valsartan
- Valsartan+Amlodipine (Experimental)
  Interventions: Drug: Amlodipine; Drug: Valsartan

INTERVENTIONS:
Drug: Amlodipine — calcium channel blocker (Amlodipine 10 mg) during 12 weeks
  Arms: Amlodipine; Valsartan+Amlodipine
Drug: Valsartan — AII receptor blocker inhibitor (Valsartan 160 mg) during 12 weeks
  Arms: Valsartan; Valsartan+Amlodipine

SUMMARY:
Diabetic nephropathy (DN) is the most important complication of diabetes mellitus (DM) and the most common cause of end-stage renal disease (ESRD). Diabetic nephropathy is a clinical syndrome characterized by persistent albuminuria (> 300 mg/d or > 200 mcg/min) that is confirmed on at least 2 occasions 3 to 6 months apart, a relentless decline in the glomerular filtration rate (GFR), and elevated arterial blood pressure. In addition to the renal hemodynamic alterations, patients with overt diabetic nephropathy (dipstick-positive proteinuria and decreasing GFR) generally develop systemic hypertension. Hypertension is an adverse factor in all progressive renal diseases and seems especially so in diabetic nephropathy. The deleterious effects of hypertension are likely directed at the vasculature and microvasculature. Use of angiotensin converting enzyme (ACE) inhibitors and/or angiotensin receptor blockers (ARBs), strict glycemic control and use of antilipidemic drugs may improve progression of DN.

TNF-like weak inducer of apoptosis (TWEAK, TNFSF12) is a member of the TNF superfamily of structurally related cytokines. The human TWEAK gene encodes a 249-amino acid type II transmembrane glycoprotein (30 kD). TWEAK may be expressed as a full-length, membrane-bound protein and as a 156-amino acid, 18-kD soluble protein, (sTWEAK) that results from proteolysis of TWEAK. TWEAK gene is expressed in many tissues, including brain, kidney, heart, arterial wall, monocytes and macrophages. Reduced soluble TNF-like weak inducer of apoptosis (sTWEAK) plasma levels have been reported both in patients with subclinical atherosclerosis and chronic kidney disease (CKD).

Long pentraxin 3 (PTX3) is a multimeric inflammatory mediator. Increased serum PTX3 levels have been reported among end-stage renal disease patients. Moreover, PTX3 has been suggested to represent a novel mortality risk factor, and elevated PTX3 levels have been shown to accompany increased albuminuria among patients with chronic kidney disease (CKD).

There is no data about the effects of Renin angiotensin system blockage (RAS), calcium channel blocker and combined drugs on TWEAK and PTX3 levels in diabetic proteinuric patients with hypertension. The aim of this study was to find out whether the beneficial effects of RAS blockage, calcium channel blocker and combined drugs in diabetic hypertensive proteinuric patients has any relation with the alteration of TWEAK and PTX3 levels. The investigators searched for the effects of angiotensin II (AII) receptor blocker (Valsartan 160 mg), calcium channel blocker (Amlodipine 10 mg) and AII receptor blocker plus calcium channel blocker (Valsartan 160 mg + Amlodipine 10 mg) on the clinical and laboratory parameters of diabetic hypertensive proteinuric patients.

DETAILED DESCRIPTION:
The patients who were non-obese (BMI<30kg/m2), non dyslipidemic (total cholesterol <200mg/dl, Triglyceride<150mg/dl), and free of cardiovascular events (negative medical history, negative ECG findings) were investigated for enrollment. CKD stage 1 patients older than 18 years of age and willing to participate to the study were screened. From the 375 patients with established type 2 diabetes mellitus+hypertension, 174 had proteinuria and/or hypertension (24 h protein excretion 1-2 g/day, systolic blood pressures ≥140mmHg and/or diastolic blood pressures ≥ 90 mmHg, respectively). All cases were first referrals and at the time of the study all were off treatment. Patients with history of coronary artery disease, smokers and those taking statins or renin-angiotensin blockers were excluded because of the effect of these factors on endothelial dysfunction. Of 174 screened patients 107 met the study criteria and were included in this study. The duration of proteinuria and diabetic nephropathy after initial diagnosis was not known.

The exclusion criteria were as follows: A)Nephrotic syndrome, B)coronary heart disease (patients with ischemic ST-T alterations and voltage criteria for LVH on electrocardiogram, and with history of revascularization or myocardial infarction), C) elevated liver enzymes (AST or ALT levels ≥ 40U/L) and D) renal failure (serum creatinine levels > 1.3 mg/dl). In order to evaluate the effect of RAS blockade on plasma TWEAK and PTX3 concentrations, patients with proteinuria were given an AII receptor blocker (Valsartan 160 mg), calcium channel blocker (Amlodipine 10 mg) and combine drug (Valsartan 160 mg + Amlodipine 10 mg) for 12 weeks. The effect of RAS blockade on insulin sensitivity and proteinuria was also investigated.

After the intervention period, blood samples were obtained for assay of plasma TWEAK and PTX3 concentrations, HbA1c , and insulin resistance scores (HOMA-IR).

Urine samples were also collected over a 24-hour period to determine the degree of proteinuria.

ELIGIBILITY:
Inclusion Criteria:

* CKD stage 1 patients
* Older than 18 years of age
* Type 2 Diabetic patients
* Proteinuria
* Hypertension

Exclusion Criteria:

* History of coronary artery disease
* Smokers
* Taking statins or renin-angiotensin blockers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2008-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Flow mediated dilatation | 12 weeks after

SECONDARY OUTCOMES:
TWEAK, PTX-3, Systolic Blood Pressure and Diastolic Blood Pressure | 12 weeks after

CONTACTS AND LOCATIONS:
Overall Officials: Mahmut Ilker Yilmaz, MD, Principal Investigator — GATA
Locations (1):
- GATA Nephrology, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Yilmaz MI, Carrero JJ, Martin-Ventura JL, Sonmez A, Saglam M, Celik T, Yaman H, Yenicesu M, Eyileten T, Moreno JA, Egido J, Blanco-Colio LM. Combined therapy with renin-angiotensin system and calcium channel blockers in type 2 diabetic hypertensive patients with proteinuria: effects on soluble TWEAK, PTX3, and flow-mediated dilation. Clin J Am Soc Nephrol. 2010 Jul;5(7):1174-81. doi: 10.2215/CJN.01110210. Epub 2010 Apr 29. PMID 20430947